CLINICAL TRIAL: NCT02351089
Title: Probiotics in Radiation-treated Gynecologic Cancer
Acronym: ProRad
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProRad
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Gastrointestinal Toxicity; Gynecologic Cancer
MeSH Terms: interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): capsules containing corn starch
  Interventions: Dietary Supplement: Capsules placebo
- Probiotic low dose (Active Comparator): capsules containing probiotic powder and corn starch
  Interventions: Dietary Supplement: Capsules probiotic powder and corn starch
- Probiotic high dose (Active Comparator): capsules containing probiotic powder and corn starch
  Interventions: Dietary Supplement: Capsules probiotic powder and corn starch

INTERVENTIONS:
Dietary Supplement: Capsules placebo — Capsules
  Arms: Placebo
Dietary Supplement: Capsules probiotic powder and corn starch
  Arms: Probiotic high dose; Probiotic low dose

SUMMARY:
The aim of the current Project is to study the efficacy of a probiotic Product in reducing the symptoms of gastrointestinal toxicity linked to the irradiation of gynecologic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with cancer in the small pelvis and waiting to receive radiotherapy either as a primary or as a secondary treatment following surgery. Chemotherapy may or may not be part of the treatment regimen.
* Age, older than 18 years old.
* Agreement for participation in the study by signed written informed consent.

Exclusion Criteria:

* Previously treated with irradiation of the pelvic area.
* Reluctance to refrain from using other probiotic products during the participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-02; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in incidence of loose/watery stools | Baseline and 10 weeks later

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Oncology, Lund, Sweden